CLINICAL TRIAL: NCT06850857
Title: Multi-Institutional Validation of the Integrated Modular Patient-Reported Outcome Assessment for Craniomaxillofacial Trauma (IMPACT)
Brief Title: Multi-Institutional IMPACT Validation
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Tennessee (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); University of Maryland (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 24-09945-XP
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Facial Injuries; Mandible Fracture; Le Fort; Zygomaticomaxillary Complex Fracture; Nasal Fracture; Orbital Fractures; Zygoma Fracture; Orbital Floor Fracture; Facial Laceration
Keywords: Facial Trauma; Maxillofacial Trauma; Patient-Reported Outcomes; Quality of Life; IMPACT; Mandible Fracture; Midface Fracture; Orbital Fracture; Nasal Fracture
MeSH Terms: conditions — Facial Injuries; Mandibular Fractures; Orbital Fractures; Zygomatic Fractures; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nasal Fractures (IMPACT-N): This group includes patients with fracture patterns that involve the nasal bones, nasal cavity, and/or sinuses, including: isolated nasal bone fractures, nasoorbitoethmoidal fractures, maxillary sinus fractures, Le Fort I-III fractures, and frontal sinus fractures.
  Interventions: Other: IMPACT-G Module; Other: IMPACT-N Module; Other: 15D Control Survey
- Orbital Fractures (IMPACT-O): This group includes patients with fracture patterns that involve the orbital walls or rim, including: isolated orbital fractures, zygomaticomaxillary complex fractures, nasoorbitoethmoidal fractures, and Le Fort II-III fractures.
  Interventions: Other: IMPACT-G Module; Other: IMPACT-O Module; Other: 15D Control Survey
- Jaw Fractures (IMPACT-J): This group includes patients with fracture patterns that involve the upper or lower jaw, including: mandible fractures, dentoalveolar fractures, and Le Fort I-III fractures. Zygomatic arch fractures will also be included given potential impairment of the jaw.
  Interventions: Other: IMPACT-G Module; Other: IMPACT-J Module; Other: 15D Control Survey

INTERVENTIONS:
Other: IMPACT-G Module — Administration of the general IMPACT survey module.
Other: IMPACT-N Module — Administration of the IMPACT-N survey module.
  Groups: Nasal Fractures (IMPACT-N)
Other: IMPACT-O Module — Administration of the IMPACT-O survey module.
  Groups: Orbital Fractures (IMPACT-O)
Other: IMPACT-J Module — Administration of the IMPACT-J survey module.
  Groups: Jaw Fractures (IMPACT-J)
Other: 15D Control Survey — Administration of the 15D QOL control survey.

SUMMARY:
The goal of this observational study is to validate a novel patient-reported outcome measure (PROM) for patients suffering maxillofacial trauma: The Integrated Modular Patient-Reported Outcome Assessment for Craniomaxillofacial Trauma (IMPACT). The primary question is:

Are the IMPACT modules valid and reliable measures to study quality-of-life (QOL) in patients with maxillofacial trauma?

Patients presenting for routine clinic follow-up for maxillofacial trauma will be invited to complete the IMPACT in addition to the 15 Dimension (15D) QOL survey as a control.

DETAILED DESCRIPTION:
Background: Maxillofacial trauma literature is dominated by objective and physician-rated outcomes, leaving a paucity of patient-reported outcome (PRO) research. In fact, no PRO measure (PROM) has ever been validated in this population, posing a tremendous barrier to our understanding of the patient experience. This project will overcome this barrier by validating a novel PROM designed by our research group: The Integrated Modular Patient-Reported Outcome Assessment for Craniomaxillofacial Trauma (IMPACT). The IMPACT is the first PROM designed for maxillofacial trauma, providing novel insight into the patient experience. In its current form, it is a 4-module survey instrument: one general module for all patients (IMPACT-G) and 3 modules specific to fractures of the nasal (IMPACT-N), orbital (IMPACT-O), and/or jaw (IMPACT-J) regions. Each module takes 2-5 minutes to complete for a total of 2-20 minutes, depending on the injury.

Objectives: This study will be a multi-institutional field test to determine the validity and reliability of using the IMPACT for measuring QOL in patients suffering maxillofacial trauma. The hypothesis is that each IMPACT module and subscale will significantly and at least moderately correlate with the 15D, an established general QOL survey instrument.

Methods: Patients with maxillofacial trauma presenting for routine follow-up within one year from their injury will be invited to complete the IMPACT and the 15D survey. Patients who completed an initial survey and return within one month will be invited to complete a second follow-up survey. The scores be tested for validity and reliability using multivariable linear regression, Pearson's r, Cronbach alpha, and test-retest reliability. The sensitivity to change and minimally clinically important difference (MCID) will also be calculated.

Impact: Validation of the first PROM for maxillofacial trauma is anticipated to have a significant and lasting impact in the field of maxillofacial trauma. This will allow researchers and clinicians to better understand the patient experience and make management recommendations accordingly. Integrating the IMPACT into future studies may revolutionize the field by providing novel evidence for controversial topics such as maxillomandibular fixation techniques, surgical approaches, adjunctive therapies, and more.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of maxillofacial trauma (fracture of any facial bone[s] and/or soft tissue injury) within 12 months of recruitment date.

Exclusion Criteria:

1. Patients presenting to clinic for reasons not related to maxillofacial trauma.
2. Patients with isolated fractures of the cranium or teeth.
3. Patients who cannot read, write, and/or speak English.
4. Patients who are unable to provide informed consent for themselves (including those who are under 18 years old, incapacitated, intoxicated, or cognitively impaired with a legal guardian)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from the population of patients presenting to clinics where facial trauma is managed, including otolaryngology, oral and maxillofacial surgery, plastic surgery, and/or ophthalmology clinic(s).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Criterion validity: Correlation of IMPACT modules with the 15D QOL control survey | When the initial survey is completed (within 12 months of the injury).
  Criterion validity will primarily be determined by calculating the correlation between each of the IMPACT module total scores and the 15D QOL control survey via Pearson's r, controlling for independent variables that influence survey scores.

SECONDARY OUTCOMES:
Reliability: Covariance of each item in the IMPACT modules and subscales | When the initial survey is completed (within 12 months of the injury).
  The reliability of each module and subscale will be measured via Cronbach alpha's measurement of internal consistency,
Sensitivity to Change: Change in IMPACT scores over the treatment course. | At the completion of the second survey.
  The sensitivity to change will be evaluated by comparing consecutive IMPACT module and subscale scores for patients who completed the survey two times.
Sensitivity to Change: Change in IMPACT scores over the treatment course. | Baseline (at recruitement, Day 0) and at 4 weeks.
  Follow-up IMPACT scores will be collected 4 weeks from the baseline recruitment and analyzed for improvement from the baseline scores.
Minimally Clinically Important Difference (MCID) | When the initial survey is completed (within 12 months of the injury).
  The MCID will be calculated for each IMPACT module and subscale via an anchor-based approach, using a single global question designed to comprehensively assess how the patient feels regarding their facial injury.

OTHER OUTCOMES:
Independent predictors of IMPACT scores | When the initial survey is completed (within 12 months of the injury).
  Independent variables that influence IMPACT scores for each module and subscale will be evaluated, including: demographics (age, sex, race, ethnicity), socioeconomic factors (social-vulnerability index, type of insurance), severity of trauma (Comprehensive facial injury [CFI] and Facial Injury Severity Score [score]), primary management (observation, closed treatment, and/or maxillomandibular fixation), multisystem trauma, and level of care (discharged from ED, admitted to floor / stepdown, or admitted to ICU).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Terwee CB, Prinsen CAC, Chiarotto A, Westerman MJ, Patrick DL, Alonso J, Bouter LM, de Vet HCW, Mokkink LB. COSMIN methodology for evaluating the content validity of patient-reported outcome measures: a Delphi study. Qual Life Res. 2018 May;27(5):1159-1170. doi: 10.1007/s11136-018-1829-0. Epub 2018 Mar 17. PMID 29550964
- [Background] Ologunde R, McLeod NMH. Use of patient-reported outcome measures in oral and maxillofacial trauma surgery: a review. Br J Oral Maxillofac Surg. 2018 Jun;56(5):371-379. doi: 10.1016/j.bjoms.2018.03.010. Epub 2018 Apr 9. PMID 29650475

DOCUMENTS (1):
  • Study Protocol (2025-06-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT06850857/Prot_001.pdf